CLINICAL TRIAL: NCT03579290
Title: A Pilot Feasibility Study of Providing Substance Use Treatment in the Black Church
Brief Title: Feasibility of Providing Computerized CBT in the Black Church
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2000022733; KL2TR001862 (NIH); 5R25DA035163-03 (NIH)
Record Dates: First submitted 2018-06-01; First posted 2018-07-06 (Actual); Results first posted 2021-02-25 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Substance Abuse
MeSH Terms: conditions — Substance-Related Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CBT4CBT program (Experimental): The 'CBT for CBT' program is modeled closely on our NIDA-published CBT manual. Seven core skill modules will cover the following topics, which correspond to the major session topics in the manual:
  Understanding and changing patterns of drug use, Coping with craving, Substance refusal skills, Seemingly irrelevant decisions, Planning for emergencies, and Problem-solving skills. Staying Safe
  Interventions: Behavioral: CBT4CBT program

INTERVENTIONS:
Behavioral: CBT4CBT program — The 'CBT for CBT' program is modeled closely on our NIDA-published CBT manual. Seven core skill modules will cover the following topics, which correspond to the major session topics in the manual:
  * Understanding and changing patterns of drug use,
  * Coping with craving,
  * Substance refusal skills,
  * Seemingly irrelevant decisions,
  * Planning for emergencies, and
  * Problem-solving skills.
  * Staying Safe

SUMMARY:
The investigator will conduct a pilot study evaluating the feasibility and acceptability of providing a computer-based program (CBT4CBT), used for the treatment of substance use disorders, in a church setting.

DETAILED DESCRIPTION:
The investigator will conduct a pilot study evaluating the feasibility and acceptability of providing a computer-based program (CBT4CBT), used for the treatment of substance use disorders, in a church setting. Forty Black adults with a current DSM-5 alcohol or substance use disorder will utilize the 'CBT for CBT' program over a period of 8 weeks. Primary outcomes will be acceptability and feasibility of providing the treatment in a church setting. If found to be acceptable and feasible, with preliminary promise for reductions in substance use, the next step would be to adapt the computer intervention for this population and conduct a randomized controlled trial.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age
* Has at least one SUD diagnosis as defined by the DSM 5

Exclusion Criteria:

* Are unable provide informed consent or participate in the study procedures as proposed in the consent
* Active suicidal or homicidal ideation
* Current engagement in substance use treatment
* Have a current legal case pending, such that incarceration during the 8 week protocol is likely
* Are in need of detoxification from alcohol, opioids or benzodiazepines

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2018-05-24 (Actual); Primary Completion 2018-10-30 (Actual); Study Completion 2018-10-30 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ayana Jordan, MD; PhD, Principal Investigator — Yale University
Locations (1):
- Dixwell Ave Congregational United Church of Christ, New Haven, Connecticut, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment occurred June through August of 2018. Participants were recruited from flyers distributed at local churches and from community services in the New Haven area. The flyers were developed with the Yale Center for Clinical Investigation (YCCI) to be culturally appropriate, and featured images of Black adults.
Groups:
- CBT4CBT Program: The 'CBT for CBT' program is modeled closely on our NIDA-published CBT manual. Seven core skill modules will cover the following topics, which correspond to the major session topics in the manual:
  Understanding and changing patterns of drug use, Coping with craving, Substance refusal skills, Seemingly irrelevant decisions, Planning for emergencies, and Problem-solving skills. Staying Safe
  CBT4CBT program: The 'CBT for CBT' program is modeled closely on our NIDA-published CBT manual. Seven core skill modules will cover the following topics, which correspond to the major session topics in the manual:
  * Understanding and changing patterns of drug use,
  * Coping with craving,
  * Substance refusal skills,
  * Seemingly irrelevant decisions,
  * Planning for emergencies, and
  * Problem-solving skills.
  * Staying Safe
Period: Overall Study
Arm/Group | CBT4CBT Program
Started | 40
Completed | 31
Not Completed | 9
Not completed — Lost to Follow-up | 9

BASELINE CHARACTERISTICS:
Arm/Group | CBT4CBT Program
Number analyzed (Participants) | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 51.9 (9.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20
  Male | 20
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 40
  White | 0
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 40
DSM 5 checklist for substance use disorders [Count of Participants; unit: Participants] — Symptoms endorsement mild 2-3 moderate (4-5) severe (6+)
  Participants
    Mild | 5
    Moderate | 13
    Severe | 22
Substance Use Calendar [Mean (Standard Deviation); unit: days] — Mean number of days of self report use of alcohol, cocaine, marijuana, opioids, benzodiazepine, heroin, nicotine for the 28 days previous to baseline.
  days
    Mean days of alcohol use past 28 days | 17.9 (10.3)
    Mean days of cocaine use past 28 days | 8.9 (11.9)
    Mean days opioid use past 28 days | 1.3 (5.0)
    Mean days of marijuana use past 28 days | 7.6 (10.6)
    Mean days of benzodiazapine use past 28 days | .31 (1.3)
    Mean days of heroin use past 28 days | 3.0 (8.0)
    Mean number of days of nicotine use past 28 days | 13.2 (13.0)
Number of Participants Testing Positive for Substance [Count of Participants; unit: Participants] — Urine toxicology screening performed by Confirm Biosciences, 12 panel, confirm insta-cup, Alcohol (EtG), Amphetamine (AMP), Barbiturates (BAR), Benzodiazepines (BZO), Cocaine (COC), Marijuana (THC), Methadone (MTD), Methamphetamine (mAMP), Ecstasy/Molly (MDMA), Opiate (OPI), Buprenorphine (BUP), Oxycodone (OXY)].
  Participants
    Number of positive for Alcohol | 16
    Number positive for Amphetamine | 1
    Number positive for Barbiturates | 2
    Number positive for Benzodiazapines | 0
    Number positive for Cocaine | 22
    Number positive for Marijuana | 16
    Number positive for Methadone | 2
    Number positive for Methamphetamine | 0
    Number positive for Ecstasy | 3
    Number positive for Opioids | 4
    Number positive for Buprenorphine | 2
    Number positive for Oxycodone | 2

OUTCOME MEASURES:

1. Primary Outcome: Recruitment Feasibility
Description: Feasibility is a composite variable (yes/no indicator). This will be determined by counting the number of participants completing the CBT4CBT intervention with significant reductions in drug use, as measured by mean change scores in the severity and quantity of substance use, and functioning over the course of treatment.
Time Frame: 8 weeks
Population: This outcome measure was never collected.
Arm/Group | CBT4CBT Program
Number analyzed (Participants) | 0

2. Primary Outcome: Program Acceptability
Description: Acceptability of treatment will be assessed by giving each participant a post-intervention satisfaction survey that assesses satisfaction with the intervention, perception of outcome, attitudes about spiritual practices accompanying CBT4CBT modules, and whether the participant would recommend this program to a friend. To evaluate the acceptability of CBT4CBT with BSUD in a church setting and to identify if religious behaviors led by trained church based health advisors (CHA), may increase the likely suitability of this intervention within the Black church.
Time Frame: 8 weeks
Population: Participants that completed the program.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | CBT4CBT Program
Number analyzed (Participants) | 31
units on a scale
  Overall Satisfaction (1-5) Very satisfied to very dissatisfied | 1.6 (0.89)
  Describe current condition at present (1-5) excellent to poor | 1.7 (.66)
  How have you changed (1-5) much worse to much better better | 3.8 (1.2)
  Are you worse, unchanged or better (1-3) | 2.6 (3.8)
  Are you better due to tx in Black Church (1-5) Definitely not related to definitely related | 3.1 (1.5)
  Satisfaction with amount of tx received (1-5) very satisfied to very dissatisfied | 1.9 (1.2)
  How satisfied were you with the CBT program (1-6) very satisfied to very dissatisfied | 1.6 (1.0)
  If seeking future tx, would you return to CBT program (1-5) Definitely to definitley not | 1.4 (.72)
  Has this tx program met your need (1-5) almost all needs to none of my needs | 2.1 (1.1)
  What will be drug and alcohol use in the next month (1-6) not use any to use daily | 2.0 (1.3)
  Able to do homework after watching example (1-5) strongly disagree to strongly agree | 3.5 (1.1)
  Homework helped me understand my drug and alcohol use (1-6) strongly disagree to strongly agree | 4.0 (1.0)
  Homework helped give me tools to help drug problem (1-6) strongly disagree to strongly agree | 4.1 (1.3)
  Satisfied with general content of CBT program (1-5) strongly dissatisfied to strongly satisfied | 3.7 (.95)
  Satisfied with ability to learn from CBT program (1-5) strongly dissatisfied to strongly satisfied | 3.7 (1.0)
  Rating for computer facilitated program as tool for learning (1-5) very poor to excellent | 3.8 (.97)

3. Primary Outcome: Sessions Attended
Description: To determine the feasibility of the program, the mean number of sessions attended was calculated per participant. The maximum number of sessions that could be attended was 7. A missed session could be made up in an additional week. The program lasted 8 weeks.
Time Frame: 8 weeks
Measure: Mean (Standard Deviation); unit: sessions
Arm/Group | CBT4CBT Program
Number analyzed (Participants) | 40
sessions | 6.8 (1.9)

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | CBT4CBT Program
All-Cause Mortality (participants affected / at risk) | 0/40
Serious Adverse Events (participants affected / at risk) | 0/40
Other Adverse Events (participants affected / at risk) | 0/40

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (3):
  • Study Protocol (2019-04-08): https://cdn.clinicaltrials.gov/large-docs/90/NCT03579290/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-03): https://cdn.clinicaltrials.gov/large-docs/90/NCT03579290/SAP_001.pdf
  • Informed Consent Form (2018-04-27): https://cdn.clinicaltrials.gov/large-docs/90/NCT03579290/ICF_002.pdf